

# Nebulised HS in children and young people with NMD or CP

A Chart Review assessing the effect of Nebulised Hypertonic Saline on Respiratory-related complications in children and young people with Neuromuscular Disease or Cerebral Palsy

Version 2, 04/04/2018

FUNDERS: This section does not apply

IRAS Project ID: 243535 REC reference: 18/YH/0103

Protocol authorised by:

Name & Role Date **Signature** 



## **Study Management Group**

Chief Investigator: Hui-Leng Tan

Co-investigators: Natalia Galaz Souza

Statistician: Mark Rosenthal

Study Management:

#### Clinical Queries

Clinical queries should be directed to Dr. Hui-Leng Tan who will direct the query to the appropriate person.

### **Sponsor**

Imperial College London is the main research Sponsor for this study. For further information regarding the sponsorship conditions, please contact the Head of Regulatory Compliance at:

Joint Research Compliance Office Imperial College London Room 215, Level 2, Medical School Building Norfolk Place London, W2 1PG

Tel: 0207 594 9459/ 0207 594 1862

http://www3.imperial.ac.uk/clinicalresearchgovernanceoffice

#### **Funder**

[This section does not apply]

This protocol describes the Nebulised Hypertonic Saline in children with Neuromuscular disease or Cerebral Palsy study and provides information about procedures for entering participants. Every care was taken in its drafting, but corrections or amendments may be necessary. These will be circulated to investigators in the study. Problems relating to this study should be referred, in the first instance, to the Chief Investigator.

This study will adhere to the principles outlined in the NHS Research Governance Framework for Health and Social Care (2<sup>nd</sup> edition). It will be conducted in compliance with the protocol, the Data Protection Act and other regulatory requirements as appropriate.

| Table of Contents | Page No |
|------------------------------------|---------|
| 1. INTRODUCTION | 6 |
| 1.1 BACKGROUND 6 | |
| 2. STUDY OBJECTIVES | 7 |
| 3. STUDY DESIGN | 7 |
| 3.1 STUDY OUTCOME MEASURES 8 | |
| 4. PARTICIPANT ENTRY | 8 |
| 4.1 PRE-REGISTRATION EVALUATIONS 8 | |
| 4.2 INCLUSION CRITERIA 8 | |
| 4.3 EXCLUSION CRITERIA 8 | |
| 4.4 WITHDRAWAL CRITERIA 8 | |
| 5. ASSESSMENT AND FOLLOW-UP | 8 |
| 6. STATISTICS AND DATA ANALYSIS | 8 |
| 7. REGULATORY ISSUES | 9 |
| 7.1 ETHICS APPROVAL 9 | |
| 7.2 CONSENT 9 | |
| 7.3 CONFIDENTIALITY9 | |
| 7.4 INDEMNITY 9 | |
| 7.5 SPONSOR 10 | |
| 7.6 FUNDING 10 | |
| 7.7 AUDITS 10 | |
| 8. STUDY MANAGEMENT | 10 |
| 9. PUBLICATION POLICY | 10 |
| 10. REFERENCES | 10 |
| APPENDICES | 13 |

## **GLOSSARY OF ABBREVIATIONS**

| AE | Adverse Event |
|--------|----------------------------------|
| CI | Chief Investigator |
| CRF | Case Report Form |
| DMC | Data Monitoring Committee |
| DOB | Date of Birth |
| GCP | Good Clinical Practice |
| HRA | Health Research Authority |
| ICF | Informed Consent Form |
| ID | Identification number |
| ISF | Investigator Site File |
| NHANES | National Health and Nutrition |
| | Examination Survey |
| PI | Principal Investigator |
| PIS | Participant Information Sheet |
| RB&HFT | Royal Brompton and Harefield NHS |
| | Foundation |
| REC | Research Ethics Committee |
| SAE | Serious Adverse Event |
| SOP | Standard Operating Procedure |
| SP | Subject Patient |
| VAS | Visual Analogue Scale |

## **KEYWORDS**

[Nebulised Hypertonic Saline, Neuromuscular disease, Cerebral Palsy, Children, Respiratory complications, Polygraphy]

#### STUDY SUMMARY





TITLE A Chart Review assesing the effects of Nebulised Hypertonic Saline on Respiratory-related complications in children and young people with Neuromuscular Disease or Cerebral Palsy

**DESIGN** Chart Review and Questionnaire application

AIMS 1)To explore whether treatment with 7% or 3% nebulised Hypertonic Saline in children and young people with Neuromuscular Disease or Cerebral Palsy decreases respiratory-related complications.

2) Assess whether the use of 3% or 7% nebulised Hypertonic Saline improves ease of airway clearance in children and young people with Neuromuscular Disease or Cerebral Palsy

#### **OUTCOME MEASURES**

- 1) Number of respiratory exacerbations requiring antibiotic treatment.
- 2) Number of hospitalisations due to respiratory exacerbations, using NHANES 2011 questionnaire for Hospitalisation and access to care HUQ.010.
- 3) Nocturnal oximetry and polygraphy outcomes: BasalSpO2 (%), Minimum SpO2 (%), Maximum SpO2 (%), Average SpO2, Oxygen desaturation index (ODI), Snoring and End tidal CO2 (EtCO2).
- 4) Rate of decline of pulmonary function.
- 5) Score on the ease of airway clearance pictorial analogue scale from participants.
- 6) Participants' perception of treatment.

#### POPULATION

Children and young people with Neuromuscular disease or Cerebral Palsy who are treated at Royal Brompton Hospital and their parents or legal guardians.

#### **ELIGIBILITY**

Inclusion cirteria: Children and young people with Neuromuscular disease or Cerebral Palsy who have their care at the Royal Brompton Hospital and are on treatment with nebulised Hypertonic Saline for at least 12 months.

Exclusion criteria: Children or young people also diagnosed with Cystic Fibrosis.

**DURATION** 6 months

#### REFERENCE DIAGRAM

[if appropriate]

#### 1. INTRODUCTION

#### 1.1 BACKGROUND

In the UK, Neuromuscular diseases have a prevalence of 118 per 100,000 people amongst adults and children. About 70% are inherited, and 13% are muscular dystrophies (1). Worldwide, the prevalence of Cerebral Palsy is 2.11 per 1000 live births (2).

The pathophysiology of neuromuscular diseases and cerebral palsy leads to restrictive pathology of the respiratory system. Children with neuromuscular diseases have several characteristics that may impair their respiratory function, such as weak bulbar and respiratory musculature, increased upper airway collapsibility and low lung compliance (3,4). Cerebral Palsy is defined as a group of disorders of the motor function, caused by a disturbance to the developing brain (5). Although pulmonary disease is not the primary diagnosis, some clinical characteristics may lead to respiratory failure. These include scoliosis, gastroesophageal reflux, and impaired swallowing, which leads to chronic aspiration, upper airway obstruction, recurrent infections, and possible bronchiectasis, developing lung disease (6). Bulbar musculature weakness impairs swallowing, which leads to chronic aspiration. Respiratory muscle weakness compromises the pump function and the effectiveness of cough. Upper airway collapsibility increases work of breathing and respiratory muscle fatigue. Low pulmonary compliance hinders the ability to expand the lung, which is exacerbated by respiratory muscle weakness, increasing the WOB. Low peak flow and decreased Vital Capacity (VC), which further decreases with progression of the disease (7), characterizes the pulmonary function of these patients. Consequently, cough may be impaired by low inspiration volumes, ineffective glottis closure and/or low expiratory force (4.8,9). Low Vital Capacity and ineffective cough in Neuromuscular disease has been associated with chronic airway inflammation and infection (9). Furthermore, children with Neuromuscular disease often have gastroesophageal reflux (GER) (10), which may cause airway inflammation (11). Chronic airway infection and colonisation of Pseudomonas aeruginosa and Gram-negative microorganisms have shown to increase morbidity of children with CP (12). GER, impaired swallowing and ineffective cough leads to chronic aspiration and contributes to recurrent pneumonias. Therefore, bronchiectasis and pulmonary fibrosis are commonly developed.

Children with Neuromuscular disease show a decline of Forced Vital Capacity (FVC), which is steeper at younger ages (13). This is especially important because the age at which FVC reaches 1 Lt and the rate of decline of FVC are variables that can predict mortality (14).

Pneumonia, respiratory exacerbations and failure are one of the most important causes of emergency admissions, hospitalisations and death in children with neuromuscular diseases and cerebral palsy (15-18). Physical health and the number of days spent outside home or hospitalised are important domains of life and predictor of Health-Related Quality of Life in children with Neuromuscular disease and children with Cerebral Palsy (19,20). In this context, it is of importance to research how to therapeutically aid airway clearance, decrease respiratory exacerbations and reduce the pulmonary function rate of decline.

Hypertonic Saline is a solution of salt water used as a nebulized medication in many conditions. Its clinical benefits include mucus clearance, microbiological diagnosis, improvement of lung function, decrease in respiratory exacerbations, cough triggering and improvement of quality of life (21). It has mucolytic and expectorant effect, reduces biofilm formation by Pseudomonas Aeruginosa and increases antioxidative thiols in the airway liquid (22).

Retrospective studies and clinical trials have shown that inhaled Hypertonic Saline is well tolerated, reduces pulmonary exacerbations, improves lung function and Lung Clearance Index, reduces absenteeism, improves Health Related Quality of Life in patients with Cystic Fibrosis independent of rhDNase treatment (23-26), and has anti-inflammatory effect in sputum decreasing



IL-8 (27). In asthmatic and healthy subjects, inhaled Hypertonic Saline have shown to enhance mucociliary clearance (28). To date, studies investigating Hypertonic Saline in bronchiectasis have produced conflicting results (29).

This study aims to assess the effectiveness of the use of nebulised Hypertonic Saline in respiratory outcomes in children and young people with Neuromuscular disease or with Cerebral Palsy.

#### 1.2 RATIONALE FOR CURRENT STUDY

[To our knowledge, there is currently no available data concerning the use of nebulised Hypertonic Saline in the management of children and young people with Neuromuscular Disease or with Cerebral Palsy. This study aims to assess whether the use of nebulised Hypertonic Saline in children and young people with Neuromuscular disease or Cerebral Palsy is effective in the management and prevention of respiratory-related complications.

Hypothesis: Nebulised Hypertonic Saline in children and young people with Neuromuscular disease or Cerebral Palsy decreases respiratory-related complications.]

#### 2. STUDY OBJECTIVES

[Primary Objective: To explore whether treatment with 3% and 7% Nebulised Hypertonic Saline in children and young people with Neuromuscular Disease or Cerebral Palsy decreases respiratory-related complications.

#### Secondary Objectives:

- Assess the effect of the treatment with nebulised hypertonic saline in children and young people with Neuromuscular disease or Cerebral Palsy on the number of courses of antibiotic prescribed compared to year before starting treatment.
- Determine whether the use of nebulised Hypertonic Saline in children and young people with Neuromuscular Disease or Cerebral Palsy reduces the frequency of hospitalisations due to respiratory exacerbations compared to year before commencing treatment.
- Explore the impact of the treatment with hypertonic saline on nocturnal oxygenation and ventilation in children and young people with Neuromuscular disease or with Cerebral Palsy.
- Evaluate whether the treatment with nebulised hypertonic saline in children and young people with neuromuscular disease or cerebral palsy improves the ease of airway clearance.
- In the subgroup of participants with neuromuscular disease who can perform spirometry, assess whether the use of Hypertonic Saline decreases rate of decline of pulmonary function compared to year before commencing treatment.
- Explore how parents of children and young people with Neuromuscular disease or with Cerebral Palsy perceive the treatment with nebulised hypertonic saline compared to previous management.

#### 3. STUDY DESIGN

[Chart review of children and young people with Neuromuscular disease or with Cerebral Palsy who are cared for in the Royal Brompton Hospital and that have been treated with nebulised hypertonic saline for at least 12 months. Children and young people who are also diagnosed with Cystic Fibrosis will be excluded.

Parents or legal guardians will be asked to complete two questionnaires to further complement data from hospital records.



Participants between 10 and 18 years old will be asked to complete one questionnaire to complement hospital records.]

[Duration: 6 months.]

[We aim to review all charts of participants recruited that meet criteria between December 2011 and May 2018. We aim to recruit 40 participants from each group, including children, young people, and parents or legal guardians, as this will be a pilot study. Only participants recruited will have their charts reviewed]

#### 3.1 STUDY OUTCOME MEASURES

**Primary Endpoints:** 

- Number of respiratory exacerbations requiring antibiotic treatment.
- Number of hospitalsiations due to respiratory exacerbations, using NHANES 2011 questionnaire for Hospitalisation and access to care HUQ.010.
- Nocturnal oximetry and polygraphy outcomes: Basal SpO2 (%), Minimum SpO2 (%), Maximum SpO2 (%), Average SpO2 (%), Oxygen desaturation index (ODI), Snoring and End tidal CO2 (EtCO2).
- Rate of decline of pulmonary function.

#### Secondary Endpoints:

- Score on the ease of airway clearance pictorial analogue scale from all participants.
- Participants' perception of treatment.

#### 4. PARTICIPANT ENTRY

#### 4.1 PRE-REGISTRATION EVALUATIONS

[This section does not apply]

#### 4.2 INCLUSION CRITERIA

[Children and young people under 18 years old with Neuromuscular disease or with Cerebral Palsy treated with nebulised Hypertonic Saline for at least 12 months and their parents or legal guardians.]

#### 4.3 EXCLUSION CRITERIA

[Children or young people who are also diagnosed with Cystic Fibrosis, as the effectiveness of nebulised Hypertonic Saline have already been studied extensively in this group.]

#### 4.4 WITHDRAWAL CRITERIA

[This section does not apply.]

#### ASSESSMENT AND FOLLOW-UP

[This section does not apply]

#### 6. STATISTICS AND DATA ANALYSIS

[Sample Size:



We aim to recruit 40 participants for each group, including children and young people and their parents or legal guardians, as this is a pilot study.

#### Statistical Analysis Plan:

Primary endpoint analysis:

- Univariate X<sup>2</sup> analysis for categorical variables to investigate *Courses of antibiotic treatment*.
- Univariate X<sup>2</sup> analysis for categorical variables to investigate *Number of hospitalisations*.
- Student t testing will be used to analyse *nocturnal oxygenation and ventilation outcomes* comparing one year before and after starting treatment with Hypertonic Saline.
- Independent t testing and Mann-Whitney U test to analyse *Rate of decline in pulmonary function*.
- Cox proportional hazard model to test differences in primary endpoints *for different baseline*

Secondary enpoint analysis:

- Univarate analysis to analyse *Ease of airway clearance*.
- Univariate analysis on **perception of treatment**.

Data and all appropriate documentation will be stored for a minimum of 10 years after the completion of the study, including the follow-up period.

#### 7. REGULATORY ISSUES

#### 7.1 ETHICS APPROVAL

The Study Coordination Centre has obtained approval from the Yorkshire & The Humber - Leeds West Research Ethics Committee (REC) and Health Regulator Authority (HRA). The study must also receive confirmation of capacity and capability from each participating NHS Trust before accepting participants into the study or any research activity is carried out. The study will be conducted in accordance with the recommendations for physicians involved in research on human subjects adopted by the 18th World Medical Assembly, Helsinki 1964 and later revisions.

#### 7.2 CONSENT

Consent to enter the study must be sought from each participant only after a full explanation has been given, an information leaflet offered, and time allowed for consideration. Signed participant consent should be obtained. The right of the participant to refuse to participate without giving reasons must be respected. After the participant has entered the study the clinician remains free to give alternative treatment to that specified in the protocol at any stage if he/she feels it is in the participant's best interest, but the reasons for doing so should be recorded. In these cases, the participants remain within the study for the purposes of follow-up and data analysis. All participants are free to withdraw at any time from the protocol treatment without giving reasons and without prejudicing further treatment.

#### 7.3 CONFIDENTIALITY

The Chief Investigator will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act.

#### 7.4 INDEMNITY

Imperial College London holds negligent harm and non-negligent harm insurance policies which apply to this study.



#### 7.5 SPONSOR

Imperial College London will act as the main Sponsor for this study. Delegated responsibilities will be assigned to the NHS trusts taking part in this study.

#### 7.6 FUNDING

This section does not apply.

#### 7.7 AUDITS

The study may be subject to inspection and audit by Imperial College London under their remit as sponsor and other regulatory bodies to ensure adherence to GCP and the NHS Research Governance Framework for Health and Social Care (2<sup>nd</sup> edition).

#### 8. STUDY MANAGEMENT

The day-to-day management of the study will be co-ordinated through Hui-Leng Tan.

#### 9. PUBLICATION POLICY

[ Data ownership rights will lie with the institution. Findings of this study will be presented as a Dissertation and will be available through Open Access. We aim to publish findings in peer-review journals. Dr. Hui-Leng Tan will take the lead in the publication and dissemination.]

#### 10. REFERENCES

- (1) Pohlschmidt M, Meadowcroft R. *Muscle disease: the impact. Incidence and Prevalence of Neuromuscular Conditions in the UK.* Muscular Dystrophy Campaign: Report number: 1, 2010.
- (2) Oskoui M, Coutinho F, Dykeman J, Jetté N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. *Developmental Medicine & Child Neurology*. 2013;55(6): 509-519.
- (3) Allen J. Pulmonary complications of neuromuscular disease: A Respiratory mechanics perspective. *Paediatric Respiratory Reviews.* 2010;11(1): 18-23. . Available from: doi: <a href="https://doi.org/10.1016/j.prrv.2009.10.002">https://doi.org/10.1016/j.prrv.2009.10.002</a>. Available from: http://www.sciencedirect.com/science/article/pii/S1526054209000700.
- (4) Lo Mauro A, Aliverti A. Physiology of respiratory disturbances in muscular dystrophies. *Breathe.* 2016;12(4): 318-327.
- (5) Rosenbaum P, Paneth NF, Leviton AF, Goldstein MF, Bax MF, Damiano DF, et al. A report: the definition and classification of cerebral palsy April 2006. *Developmental medicine and child neurology.Supplement JID 0006762.* 2007;1098-14.
- (6) Fitzgerald DA, Follett J, Van Asperen PP. Assessing and managing lung disease and sleep disordered breathing in children with cerebral palsy. *Paediatric Respiratory Reviews.* 2009;10(1): 18-24. . Available from: doi: <a href="https://doi.org/10.1016/j.prrv.2008.10.003">https://doi.org/10.1016/j.prrv.2008.10.003</a>. Available from: http://www.sciencedirect.com/science/article/pii/S1526054208000729.

- (7) Bushby K, Finkel R, Birnkrant DJ, Case LE, Clemens PR, Cripe L, et al. Diagnosis and management of Duchenne muscular dystrophy, part 1: diagnosis, and pharmacological and psychosocial management. *The Lancet Neurology*. 2010;9(1): 77-93.
- (8) Boitano LJ. Management of Airway Clearance in Neuromuscular Disease. *Respiratory care*. 2012;51(8): 913-924. . Available from: <a href="http://rc.rcjournal.com/content/51/8/913.abstract">http://rc.rcjournal.com/content/51/8/913.abstract</a>.
- (9) Stehling F, Pieper N, Bouikidis A, Steinmann J, Rath P, Mellies U. Upper airway microbial colonization in patients with neuromuscular disorders. *Respirology*. 2016;21(7): 1285-1291.
- (10) Skalsky AJ, Dalal PB. Common Complications of Pediatric Neuromuscular Disorders. *Physical Medicine and Rehabilitation Clinics of North America.* 2015;26(1): 21-28. . Available from: doi: <a href="https://doi.org/10.1016/j.pmr.2014.09.009">https://doi.org/10.1016/j.pmr.2014.09.009</a> ". Available from: <a href="http://www.sciencedirect.com/science/article/pii/S1047965114001065">http://www.sciencedirect.com/science/article/pii/S1047965114001065</a>.
- (11) Carpagnano GE, Resta O FAU Ventura,,M.T., FAU VM, FAU AA, Di Gioia GF, Giliberti TF, et al. Airway inflammation in subjects with gastro-oesophageal reflux and gastro-oesophageal reflux-related asthma. *Journal of internal medicine*. 2006;259(3): 323-331.
- (12) Gerdung CA, Tsang A, Yasseen AS, Armstrong K, McMillan HJ, Kovesi T. Association Between Chronic Aspiration and Chronic Airway Infection with Pseudomonas aeruginosa and Other Gram-Negative Bacteria in Children with Cerebral Palsy. *Lung.* 2016;194(2): 307-314.
- (13) Kohler M, Clarenbach CF, Böni L, Brack T, Russi EW, Bloch KE. Quality of Life, Physical Disability, and Respiratory Impairment in Duchenne Muscular Dystrophy. *Am J Respir Crit Care Med.* 2005;172(8): 1032-1036.
- (14) Phillips MF, Quinlivan RCM, Edwards R , Calverley PM . Changes in Spirometry Over Time as a Prognostic Marker in Patients with Duchenne Muscular Dystrophy. *Am J Respir Crit Care Med.* 2001;164(12): 2191-2194.
- (15) Bell CF, Kurosky SK, Candrilli SD. Muscular dystrophy-related hospitalizations among male pediatric patients in the United States. *Hospital practice*. 2015;43(3): 180-185.
- (16) Van Ruiten HJA, Marini Bettolo C, Cheetham T, Eagle M, Lochmuller H, Straub V, et al. Why are some patients with Duchenne muscular dystrophy dying young: An analysis of causes of death in North East England. *European Journal of Paediatric Neurology.* 2016;20(6): 904-909. Available from: doi: <a href="https://doi.org/10.1016/j.ejpn.2016.07.020">https://doi.org/10.1016/j.ejpn.2016.07.020</a>. Available from: <a href="https://www.sciencedirect.com/science/article/pii/S109037981630126X">https://www.sciencedirect.com/science/article/pii/S109037981630126X</a>.
- (17) Meehan E, Reid SM, Williams K, Freed GL, Sewell JR, Vidmar S, et al. Hospital admissions in children with cerebral palsy: a data linkage study. *Developmental medicine and child neurology*. 2017;59(5): 512-519.
- (18) Meehan E, Reid SM, Williams K, Freed GL, Babl FE, Sewell JR, et al. Tertiary paediatric emergency department use in children and young people with cerebral palsy. *Journal of paediatrics and child health.* 2015;51(10): 994-1000.

- (19) Davis E, Reddihough D, Murphy N, Epstein A, Reid SM, Whitehouse A, et al. Exploring quality of life of children with cerebral palsy and intellectual disability: What are the important domains of life? *Child: Care, Health and Development.* 2017;43(6): 854-860.
- (20) Otto C, Steffensen BF, Højberg A, Barkmann C, Rahbek J, Ravens-Sieberer U, et al. Predictors of Health-Related Quality of Life in boys with Duchenne muscular dystrophy from six European countries. *Journal of neurology*. 2017;264(4): 709-723.
- (21) Rogers DF. Mucoactive agents for airway mucus hypersecretory diseases. *Respiratory care:* the official journal of the American Association for Respiratory Therapy. 2007;52(9): 1176-1197.
- (22) Elkins MR, Bye PT. Mechanisms and applications of hypertonic saline. *J R Soc Med.* 2011;104(1): 2-5.
- (23) Dmello D, Nayak RP, Matuschak GM. Stratified assessment of the role of inhaled hypertonic saline in reducing cystic fibrosis pulmonary exacerbations: a retrospective analysis. *BMJ Open.* 2011;1(1): 1-4. . Available from: doi: 10.1136/bmjopen-2010-000019. Available from: http://bmjopen.bmj.com/content/1/1/e000019.
- (24) Elkins MR, Robinson M, Rose BR, Harbour C, Moriarty CP, Marks GB, et al. A Controlled Trial of Long-Term Inhaled Hypertonic Saline in Patients with Cystic Fibrosis. *N Engl J Med.* 2006;354(3): 229-240.
- (25) Amin R, Subbarao P, Jabar A, Balkovec S, Jensen R, Kerrigan S, et al. Hypertonic saline improves the LCI in paediatric patients with CF with normal lung function. *Thorax.* 2010;65(5): 379-383. . Available from: doi: 10.1136/thx.2009.125831. Available from: http://thorax.bmj.com/content/65/5/379.abstract.
- (26) Donaldson SH, Bennett WD, Zeman KL, Knowles MR, Tarran R, Boucher RC. Mucus clearance and lung function in cystic fibrosis with hypertonic saline. *The New England journal of medicine*. 2006;354241-250.
- (27) Reeves EP, Williamson M, O'Neill SJ, Greally P, McElvaney NG. Nebulized Hypertonic Saline Decreases IL-8 in Sputum of Patients with Cystic Fibrosis. *Am J Respir Crit Care Med.* 2011;183(11): 1517-1523.
- (28) Daviskas E, Anderson S, Gonda I, Eberl S, Meikle S, Seale J, et al. Inhalation of hypertonic saline aerosol enhances mucociliary clearance in asthmatic and healthy subjects. *European Respiratory Journal*. 1996;9(4): 725-732. Available from: <a href="http://erj.ersjournals.com/content/9/4/725.abstract">http://erj.ersjournals.com/content/9/4/725.abstract</a>.
- (29) Hart A, Sugumar K FAU Milan, Stephen, J., FAU MS, FAU FS, Crossingham I. Inhaled hyperosmolar agents for bronchiectasis. *The Cochrane database of systematic reviews JID 100909747.* 1996;9(4): 725-732.



#### **APPENDICES**

- Appendix 1 Questionnaire on Hypertonic Saline treatment for parents and legal guardians.
- **Appendix 2** Questionnaire on Hypertonic Saline treatment for participants 16 18 years.
- **Appendix 3** Questionnaire on Hypertonic Saline treatment for participants 10 15 years.
- Appendix 4 Consent form
- Appendix 5 Consent form
- Appendix 6 Assent form

# Hypertonic saline treatment questionnaire PARENTS/LEGAL GUARDIAN

| Participant II | D: | | | | | | | | Date: | / | / |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1)Overall, d<br>had has bee | | eel th | at neb | ulised | hypert | onic sa | line yo | ur child | l / your | ng perso | n has |
| | ul<br>useful<br>n't know | , | | | | | | | | | |
| What have yo | u found | most ( | useful a | bout it? | • | | | | | | |
| What have yo | u found | most o | difficult, | / trouble | esome a | bout it? | | | | | |
| 2)Please sco<br>airway<br>Before startin | | | | ink it l | nas bee | n to cle | ear spu | tum fro | om your | child's | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| | + | + | $\dashv$ | + | $\dashv$ | + | $\dashv$ | + | + | $\dashv$ | |
| Most Easy | | <u> </u> | | | | | | | · • • | ► Most D | ifficult |
| After starting | Hyperto | nic Sal | ine | | | | | | | | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| 1 | 1 | 1 | - 1 | - 1 | - 1 | - 1 | - 1 | - 1 | - 1 | 1 | |
| | $\top$ | $\top$ | | | | | | | | $\dashv$ | |
| Most Fasy | | | | | | | | | | Most D | ifficult |

| Participant ID: | | Date:/ |
|---|---|---|
| In the 12 months <u>before</u> starting did your child need? If you don't | | |
| Oral | | |
| IV | | |
| In the 12 months <u>after</u> starting H<br>your child need? If you don't rem | · | urses of antibiotics did |
| Oral | | |
| IV | | |
| In the 12 months <u>before</u> starting<br>take your child to see a doctor be<br>don't remember, please leave it b | ecause s/he was unwell with a | |
| In the 12 months <u>after</u> starting<br>take your child to be seen by a do<br>If you don't remember, please lea | octor because s/he was unwell | |

# Hypertonic saline questionnaire

Ages 16 to 18 years

| Participant ID: | Date: | _/ | _/ |
|---|---|---|---|
| 1)Overall, do you feel that nebulised hypertonic saline has been | | | |
| Useful<br>Not useful<br>I don't know | | | |
| What have you found most useful about it? | | | |

What have you found most difficult/ troublesome about it?

#### 2)Please score your perception of how easy it is to clear sputum.

Before starting Hypertonic Saline



After starting Hypertonic Saline



# Hypertonic saline questionnaire

AGES 10 to 15 YEARS

| Participant ID: | Date:/ |
|---|---|
| 1) Do you feel that nebulised hypertonic saline has been | |
| Useful<br>Not useful<br>I don't know | |
| What do you like about it? | What do you not like about it? |

2) Please point on the line below, between EXTREMELY EASY and EXTREMELY HARD, to show how easy it is to clear your sputum.

Before starting Hypertonic Saline



After starting Hypertonic Saline





Joint Research Compliance Office

# Imperial College London

Imperial College London

St Mary's Campus Praed St., Paddington, London W2 1NY Tel: +44 02033126666

www.imperial.ac.uk

A Chart Review assessing the effect of Nebulised Hypertonic Saline on Respiratory-related complications in children and young people with Neuromuscular Disease or Cerebral Palsy

IRAS Project ID: 243535

| | INAS FTOJECT | ID. 243333 |
|---|---|---|
| | CONSENT FORM | |
| | (16 - 18 years) | |
| | articipant Identification Number for this trial: ame of Researcher: | |
| | Please initial box if | you agree |
| 1. | I confirm that I have read and understood the information sheet version n°2 date 04/04/2018, for the above study. I have had the opportunity to consider the information, ask questions and have these answered satisfactorily. | |
| 2. | I understand that participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | |
| 3. | 3. I understand that the study research team will review relevant sections of my medical records and data. | |
| 4. I understand that data collected during the study may be looked at by responsible individuals, from regulatory authorities, Imperial College London or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | |
| 5. | I agree to fill in the study questionnaires. | |
| 6. | I agree to my parents completing the study questionnaires. | |
| Na | ame of Participant Date Signature | _ |
| Na | ame of Person taking consent Date Signature | |
| W | /hen completed, 1 for participant; 1 for researcher site file; 1 (original) to be kept in me | dical notes |



Joint Research Compliance Office

# Imperial College London

Imperial College London

St Mary's Campus
Praed St., Paddington, London
W2 1NY

Tel: +44 02033126666 www.imperial.ac.uk

A Chart Review assessing the effect of Nebulised Hypertonic Saline on Respiratory-related complications in children and young people with Neuromuscular Disease or Cerebral Palsy

IRAS Project ID: 243535

| | | CONSENT FORM | Л | |
|---|---|---|---|---|
| | pant Identification Number | er for this trial: | | |
| Name | of Researcher: | | | |
| | | | Please initial box if | you agree |
| 1. | I confirm that I have read and understood the information sheet version n°2 date 04/04/2018, for the above study. I have had the opportunity to consider the information, ask questions and have these answered satisfactorily. | | | |
| 2. | I understand that participation is voluntary and that I am free to withdraw my child at any time, without giving any reason, without affecting my child's medical care or legal rights being affected. | | | |
| 3. | <ul> <li>I understand that the study research team will review relevant sections of my<br/>child's medical records and data.</li> </ul> | | | |
| 4. | I understand that data collected during the study may be looked at by responsible individuals, from regulatory authorities, Imperial College London or from the NHS Trust, where it is relevant to my child taking part in this research. I give permission for these individuals to have access to my child's records. | | | |
| 5. | 5. I agree to my child completing the study questionnaire. | | | |
| Name | of Parent | Date | Signature | _ |
| Name of Participant | | Date | Signature (if appropriat | e) |
| Name | of Person taking consent | Date | Signature | _ |
| When | completed 1 for participa | ant: 1 for researcher site fi | le: 1 (original) to be kent in me | dical notes |



Joint Research Compliance Office

# Imperial College London

Imperial College London

St Mary's Campus Praed St., Paddington, London W2 1NY

Tel: +44 02033126666

www.imperial.ac.uk

A Chart Review assessing the effect of Nebulised Hypertonic Saline on Respiratory-related complications in children and young people with Neuromuscular Disease or Cerebral Palsy

IRAS Project ID: 243535

| | INFORMED ASSENT FORM | | | |
|---|---|---|---|---|
| Partici<br>Name | Please circle all that ye | ou | | |
| agree<br>1. | gree <ol> <li>Do you understand what this study is about?</li> </ol> | | | |
| 2. | Have you asked all the ques | tions you want? | • | Yes/No |
| 3. | . Have you had your questions answered in a way you understand? | | | |
| 4. Do you want to take part? | | | | |
| If any | answer is "No", don't sign | your name. | | |
| Name | of Participant | Date | Signature | |
| Name | of Person taking assent | Date | Signature | _ |
| When | When completed, 1 for participant; 1 for researcher site file; 1 (original) to be kept in medical notes | | | |